CLINICAL TRIAL: NCT05411679
Title: A Phase 2 Multi-arm, Open Label Study to Assess the Safety and Efficacy of EP0057 in Combination With Olaparib in Defined Populations of Patients With Relapsed Advanced Gastric Cancer and Small Cell Lung Cancer
Brief Title: EP0057 in Combination With Olaparib in Relapsed Advanced Gastric Cancer and Small Cell Lung Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Futility analysis decision to terminate EP0057 compound and all Ellipses sponsored studies involving EP0057.
Sponsor: Ellipses Pharma (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EP0057-202
Record Dates: First submitted 2022-05-25; First posted 2022-06-09 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Gastric Cancer; Small-cell Lung Cancer
Keywords: ATM-negative gastric cancer
MeSH Terms: conditions — Stomach Neoplasms; Small Cell Lung Carcinoma | interventions — olaparib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm 1 (Experimental): patients with ataxia-telangiectasia mutated protein (ATM)-negative relapsed, advanced GC.
  Interventions: Drug: EP0057; Drug: Olaparib tablets
- Arm 2 (Experimental): patients with relapsed extensive stage SCLC.
  Interventions: Drug: EP0057; Drug: Olaparib tablets

INTERVENTIONS:
Drug: EP0057 — EP0057 is an investigational nanoparticle-drug conjugate with a Camptothecin payload, that is administered intravenously
Drug: Olaparib tablets — Olaparib is a PARP inhibitor (poly [adenosine diphosphate-ribose] polymerase inhibitor) Other names: Lynparza

SUMMARY:
The aim of EP0057 - 202 is to assess the safety and efficacy of EP0057 in combination with Olaparib (a PARP inhibitor) in two cancers where there is a high unmet need: extensive stage small cell lung cancer (SCLC) and ATM-negative gastric cancer (GC).

EP0057-202 is a non-comparative, multi-arm, multi-centre, open label, Phase 2 study to determine the efficacy, safety, and tolerability of EP0057 in combination with olaparib (an approved PARP inhibitor) in defined patient populations with relapsed* GC and SCLC.

*(see Eligibility Criteria for definition of "relapse" for each tumour type/population) The treatment cohorts will open sequentially at the Sponsor's discretion and patients may be enrolled into each cohort concurrently.

EP0057 is an investigational nanoparticle-drug conjugate administered intravenously. The rationale for developing EP0057 is to enable selective entry of EP0057 into tumour tissue and as a result create preferential accumulation of EP0057, and therefore of the payload Camptothecin, to translate into maximum tumour cell killing.

DETAILED DESCRIPTION:
EP0057 - 202 is a Phase 2 multi arm, open label study in defined populations of patients with SCLC and GC.

The Primary objectives of Arm 1 will be to investigate the efficacy, as defined by best Objective Response Rate (ORR) of EP0057 in combination with Olaparib in patients with ataxia-telangiectasia mutated protein (ATM)-negative relapsed, advanced GC.

The Primary objectives of Arm 2 will be to investigate the efficacy, as defined by the best ORR of EP0057 in combination with Olaparib in patients with relapsed extensive stage SCLC.

The secondary objectives of both arms will be to further investigate the efficacy of EP0057 in combination with olaparib in the target patient population of each arm by assessment of the following:

* Progression-free survival (PFS)
* Overall survival (OS)
* Duration of overall response (DoR)
* Disease control rate (DCR)

Secondary objectives of arms 1 and 2 also include exploring the safety and tolerability of EP0057 when combined with olaparib in patients with GC and SCLC.

Exploratory objectives may or may not be performed during the course of the study, but if so, where available at the time of publication, results from these analyses will be reported in the clinical study report (CSR). Exploratory objectives are to:

* Examine the PK characteristics of EP0057 in combination with olaparib
* Investigate the impact of HRD (homologous recombination deficiency) status on primary and secondary endpoints, as analysed by sub-groups of HRD status.

It is estimated that approximately 115 patients will be enrolled into the study. The study will aim to recruit 34 patients across both arms of the study in stage 1. The study will then aim to recruit an additional 81 patients across both arms in the second stage.

ELIGIBILITY:
Inclusion Criteria:

Applicable to both arms:

1. Patients aged≥ 18 years (or legal age of majority in the jurisdiction) of age at the time of informed consent
2. Ability to understand and provide written informed consent prior to undergoing any study procedures
3. Life expectancy of > 3 months, as estimated by the Investigator
4. Presence of at least 1 measurable lesion using CT/MRI as defined by RECIST v1.1
5. Adequate haematological and organ function

   * Haemoglobin ≥9.0 g/dL
   * ANC ≥1.5 x 10^9/L
   * Lymphocyte count ≥0.5 x 10^9/L
   * Platelet count ≥100 x 10^9/L
   * Total bilirubin ≤1.5 institutional ULN
   * Serum albumin ≥2.5 g/dL
   * Aspartate transaminase (AST)and alanine transaminase (ALT) ≤2.5 x ULN, unless liver metastases are present in which case, they must be ≤5xULN
   * Creatinine clearance >50 mL/min (calculated using the Cockcroft-Gault formula) for patients with creatinine levels above institutional normal
   * Patients not receiving anti-coagulant medication must have an INR of ≤1.5 and an aPTT ≤1.5xULN
6. In the opinion of the Investigator, all other relevant medical conditions must be well-managed and stable for ≥28days prior to first administration of study drug
7. Willing and able to participate in all required evaluations and procedures in this study protocol
8. Contraception:

   For female subjects: each female subject of childbearing potential must agree to use two highly effective methods of contraception (ie, a method with less than 1% failure rate per year [eg, sterilization, hormone implants, hormone injections, some intrauterine devices, vasectomized partner, or combined birth control pills]) from screening until 6 months after the last dose of EP0057 or olaparib, whichever was taken last. Females of childbearing potential must have a negative serum pregnancy test at Screening and a negative serum or urine pregnancy test within 24 hours before each dose of EP0057 (and must not be lactating). Each female subject will be considered to be of childbearing potential unless she has been surgically sterilized by hysterectomy or bilateral tubal ligation/salpingectomy or has been postmenopausal for ≥1 year. For male subjects: Sexually active male patients must be willing to use barrier contraception (ie, condoms with spermicide) with all sexual partners for the duration of the study and for 6months after the last EP0057 administration. Where a sexual partner of a male participant is a 'woman of child-bearing potential', she must use a highly effective method contraceptive measures (see above definition) during her partner's participation in the study and for 6 months after her partner has received his last dose of EP0057. Men must not donate sperm for 6 months after the last dose of EP0057.
9. ECOG Performance Status Grade 0-2

   Arm 1 (ATM-negative relapsed advanced GC) Specific Inclusion Criteria:

   Patients must meet all of Arm 1-specific Inclusion Criteria and all of the Inclusion Criteria applicable to both arms to be eligible for inclusion in the study:
10. Confirmed histological (cytological diagnosis excluded) of gastric adenocarcinoma or gastro-oesophageal junction adenocarcinoma with archival tumour sample available. In the absence of an archival tumour biopsy sample, a tumour biopsy will need to be collected
11. HER2status known with no HER2 expression.PDL-1 status known (this does not need to be known prior to enrolment)
12. ATM protein expression known by investigational use only immunohistochemical Ventana ATM (Y170) assay, with ATM-negative status confirmed (defined as <25% nuclear staining)
13. Relapse, defined as: clear, documented evidence of locally advanced or metastatic, unresectable disease progression following: -two prior lines of systemic therapy, providing patients have not received irinotecan in the second line setting OR One prior line of therapy if considered to be unwilling or unsuitable for current standard of care treatment options

    Arm2 (Relapsed, extensive stage SCLC) Specific Inclusion Criteria:

    Patients must meet all of Arm 2-specific Inclusion Criteria and all of the Inclusion Criteria applicable to both arms to be eligible for inclusion in the study
14. Confirmed histological (cytological diagnosis excluded) SCLC with archival tumour sample available. In the absence of an archival tumour biopsy sample, a tumour biopsy will need to be collected. Note: Patients are eligible irrespective of prior assessment of limited or extensive disease
15. PDL-1 status known (this does not need to be known prior to enrolment)
16. Relapse, defined as: clear, documented evidence of disease progression following at least one (and no more than two) lines of previous therapy. Patients must have received all available standard of care treatment options or be unsuitable or unwilling to receive the current standard of care treatment

Exclusion Criteria:

* Applicable to both arms:

  1. Unresolved or unstable serious toxic side-effects of prior chemotherapy or radiotherapy, ie, Grade≥2 per CTCAE (v5.0) except fatigue, alopecia, infertility, or palliative radiotherapy within 6 weeks prior to start of study treatment
  2. Known cerebral metastases or CNS involvement including leptomeningeal disease. SCLC patients should not have imaging older than 2 weeks prior to start of screening to exclude brain disease. For GC patients, imaging should not be older than 12 weeks prior to start of screening to exclude brain disease. Note: Any abnormal findings on brain imaging should be discussed with the Medical Monitor as part of the screening process

     • Subjects with previously treated brain metastases are eligible to participate if: a) they are stable (no evidence of progression by imaging; same imaging modality [MRI or computed tomography (CT) scan] must be used for each assessment) for at least 28 days prior to the first dose of study drug; b) any neurologic symptoms returned to baseline; c) they have no evidence of new or enlarging brain metastases; d) they are not using corticosteroids for at least 7 days prior to the first dose of study drug.
  3. Malignant disease other than that being treated in this study, with the following exceptions:

     * Malignancies that were treated curatively and have not recurred within 2 years prior to study treatment
     * Completely resected basal cell and squamous cell skin cancers
     * Any malignancy considered to be indolent and that has never required therapy
     * Completely resected carcinoma in situ of any type
  4. Concurrent treatment with other systemic anti-cancer therapy or investigational anti-cancer drugs within 3 weeks (or 5 half-lives, whichever is longer), or 4 weeks for immunotherapy, prior to the start of study treatment
  5. Prior treatment with a topoisomerase I inhibitor
  6. History of stroke, transient ischemic attack, or myocardial infarction, within 6 months prior to C1D1
  7. Uncontrolled pleural effusion, pericardial effusion or ascites requiring recurrent drainage procedures (as defined as once monthly or more frequently). N. B - patients with indwelling catheters (eg, PleurX) are allowed
  8. Confirmed QTcF > 470 ms on screening ECG or history of Torsades de pointes or history of congenital long QT syndrome
  9. Any evidence of severe or uncontrolled systemic conditions (eg, severe hepatic impairment) or current unstable or uncompensated respiratory or cardiac conditions which makes it undesirable for the patient to participate in the study or which could jeopardize compliance with the protocol
  10. Any other concurrent severe and/or uncontrolled medical or surgical condition which, in the view of the Investigator, could compromise the patient's participation in the study
  11. Patients with active hepatitis infection (defined as having a positive HBsAg test at screening) or hepatitis C. Patients with past HBV infection or resolved HBV infection (defined as having a negative HBsAg test and a positive antibody to hepatitis B core antigen [anti-HBc], and surface antigen [anti-HBs] antibody test and no HBV DNA detectable without HBV therapy) are eligible. Patients positive for HCV antibody are eligible only if polymerase chain reaction is negative for HCV RNA
  12. Active infection with SARS-Cov-2. All patients should be tested for active SARS-Cov-2 infection with an approved diagnostic kit
  13. Patients with active HIV infection or known history of HIV infection
  14. Active infection requiring IV antibiotics within two weeks prior to treatment
  15. Women who are pregnant, likely to become pregnant, breast-feeding or either unable to or refuse to use effective means of contraception during treatment
  16. Any major surgical procedure (planned or anticipated) (in the Investigator's judgement) within 2weeks of the first dose of study treatment
  17. Known contra-indications, hypersensitivity, or severe intolerance to topoisomerase I inhibitors or Olaparib or the excipients of EP0057 or olaparib
  18. Patients with a history, or features suggestive, of bone marrow dysplasia, MDS, or AML
  19. The patient is unable to swallow capsules and/or has a surgical or anatomical condition that precludes swallowing and absorbing oral medication on an ongoing basis
  20. Concurrent treatment with potent inhibitors or inducers of CYP3A4.
  21. Concurrent treatment with Coumadin (Warfarin)
  22. Patients considered by the Investigator to be at a higher baseline risk for new onset cystitis (see Section 7.5.4)
  23. Palliative radiotherapy (e.g., for pain or bleeding) within 6 weeks prior to enrolment or patients who have not completely recovered (Grade ≥ 2) from the effects of previous radiotherapy
  24. Any other condition that would, in the Investigator's judgement, contraindicate the patient's participation in the clinical study due to safety concerns or compliance with clinical study procedures or interpretation of study results

      Arm 1 (ATM-negative relapsed advanced GC) Specific Exclusion Criteria:
  25. Prior irinotecan in the second line setting

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-04 (Estimated); Primary Completion 2024-08 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) as measured using RECIST v1.1 | Approximately 18 months

SECONDARY OUTCOMES:
Progression Free Survival (PFS) as measured using RECIST v1.1 | Approximately 18 months
Duration of Overall Response (DoR) as measured using RECIST v1.1 | Approximately 18 months
Disease Control Rate (DCR) as measured using RECIST v1.1 | Approximately 18 months
Overall Survival (OS) defined as time from start of study treatment until date of death due to any cause | Approximately 18 months
Incidence of treatment emergent adverse events (AE's) as assessed by NCI CTCAE version 5 | Approximately 18 months
Incidence of treatment emergent serious adverse events (SAE's) | Approximately 18 months
Incidence of treatment-emergent Grade ≥ 3 AEs | Approximately 18 months
Incidence of treatment-emergent AEs leading to discontinuation of trial therapy | Approximately 18 months
Incidence of treatment-emergent AEs leading to interruption of trial therapy | Approximately 18 months
Incidence of treatment-emergent AEs leading to dose reduction of trial treatment | Approximately 18 months

OTHER OUTCOMES:
Plasma levels of total and free CPT | Approximately 18 months
  Derived PK parameters will include: Cmax
Plasma levels of total and free CPT | Approximately 18 months
  Derived PK parameters will include: tmax
Plasma levels of total and free CPT | Approximately 18 months
  Derived PK parameters will include: t½
Plasma levels of total and free CPT | Approximately 18 months
  Derived PK parameters will include: AUC0-48 for C1D1 dosing
HRD status of patients | Approximately 18 months
Duration of CFT following first-line chemotherapy prior to subsequent progression | Approximately 18 months
Magnitude of response to first-line chemotherapy | Approximately 18 months

CONTACTS AND LOCATIONS:
Locations (21):
- China (8):
  - Shanghai Chest Hospital, Shanghai, Changning District, 交通大学 邮政编码
  - Fudan University Shanghai Cancer Center, Shanghai, Dongan Rd, 270, Xuhui District
  - Henan Cancer Hospital, Henan, Jinshui District, Zhengzhou
  - Linyi Cancer Hospital, Linyi, Linyi, Lanshan District, Shandong
  - The First Affiliated Hospital of Xiamen University, Fujian, Siming District, Xiamen
  - Hunan Cancer Hospital & The Affiliated Cancer Hospital of Xiangya School of Medicine, Central South, Changsha, Tongzipo Road, Yuelu District
  - Shanxi Cancer Hospital, Shanxi, Xinghualing District, Taiyuan
  - Affiliated Hospital of Hebei University, Baoding, Yuhua East Road 212, Lianchi District
- South Korea (8):
  - Seoul St. Mary Hospital, Seoul, Banpo-daero 222, Banpo-dong, Seocho-gu
  - Dong-A University Hospital, Busan, Daesingongwon-ro 26, Seo-gu
  - Seoul National University Bundang Hospital, Seoul, Gumi-ro 82 173(baekchilsipsam)beo, Bundang-gu, Seongnam-si
  - Samsung Medical Center, Seoul, Irwon-ro 81, Gangnam-gu
  - South Korea University Hospital, Seoul, Jongno-gu, Daehak-ro, 101
  - Asan Medical Center, Seoul, Olympic-ro 88 43-gil, Songpa-gu
  - Chungbuk National University Hospital, Cheongju-si, Sunhuanro 776 (1), Heungduk-gu, Cheongju-city
  - Cha University Bundang Medical Center, Gyeonggi-do, Yatap-ro 59, Bundang-gu, Seongnam
- Taiwan (5):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City, No. 100號, Ziyou 1st Rd, Sanmin District
  - Changhua Christian Hospital, Changhua, No. 176, Zhonghua Rd
  - Tapei Medical University - Shuang-Ho Hospital Ministry of Health and Welfare, New Taipei City, No. 291, Zhongzheng Rd, Zhonghe District
  - Chang Gung Medical Foundation Linkou, Taoyuan District, No.5, Fuxing St., Guishan Dist
  - Chi Mei Hospital Liouying, Tainan, Yongkang District, Zhonghua Rd, 710